CLINICAL TRIAL: NCT01318213
Title: Effect of the Use of Universal Glove and Gowning on Healthcare Associated Infection Rates and Antibiotic Resistant Bacteria
Brief Title: Benefits of Universal Glove and Gowning
Acronym: BUGG
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Centers for Disease Control and Prevention (U.S. Federal Agency); University of Iowa (Other); Joint Commission on Accreditation of Healthcare Organizations (Other)
Responsible Party: Principal Investigator, Anthony Harris, Professor, University of Maryland, Baltimore
Other Study IDs: HP-00047673; HHSA290200600015i (Other Grant/Funding Number: AHRQ PRISM No. HHSA29032002T)
Record Dates: First submitted 2011-03-16; First posted 2011-03-18 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: MRSA; VRE
Keywords: VRE; MRSA

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasal and peri-rectal culture samples will be banked in the research laboratory of Dr. J. Kristie Johnson at the University of Maryland, School of Medicine. The samples will be labeled with a participant ID without any personal identifiers. The entire sample will not be used for this study. The remaining samples will be used for future research to answer any infection control questions that arise about infection control in intensive care units that may be answered with these samples. The remaining samples will be frozen and stored indefinitely. The freezing method that will allow the study of other bacteria has been validated. Depending upon the results, there may be some rationale for thawing the samples and processing them for other antibiotic-resistant bacteria
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Intervention Arm: The intervention will consist of wearing gloves and gowns for all patient contact in the ICUs that are randomized to receive the intervention. During the intervention phases of the study, all healthcare workers (nurses, physicians, nurse extenders, respiratory therapists, social workers etc.) in the intervention group will be required to wear gloves and gowns for patient contact and when entering any patient room. In essence, healthcare workers will apply the CDC Contact Precautions guidelines for ALL patients.
- Non-intervention - Usual Standard of Care: The non-intervention units will follow their present standard of care. For all of these units, this will consist of healthcare workers following Contact Precautions (gloves and gowns) only for patients known to have antibiotic-resistant bacteria such as VRE and MRSA based on previous admission clinical and surveillance cultures or clinical cultures from the present admission. This represents on average 20-25% of patients on Contact Precautions. For the rest of the patients standard precautions will be followed.

SUMMARY:
This study will test if doctors, nurses and other people who take care of patients in hospitals wearing gloves and gown for all contact with patients in an intensive care unit (ICU) will:

* Decrease the chance of patients getting an infection while in the hospital
* Decrease the chance of patients picking up bacteria as a result of being in the hospital
* Decrease the time a patient spends in the ICU or in the hospital
* Increase the frequency of adverse events

The study will also look at whether making doctors, nurses and other people who take care of patients wear gloves and gown for all contact with patients will decrease the amount of time healthcare workers spend with patients.

This study will gather information by comparing what happens in ICUs that continue to do what they were doing before the study with what happens in ICUs that require healthcare workers to wear gloves and gown for all contact with patients.

This study will provide information that will help to make being in the hospital safer for all patients.

DETAILED DESCRIPTION:
GOAL:

The overall goal of this project is to determine the effectiveness of universal glove and gowning procedures in reducing healthcare-associated infection (HAI) rates and acquisition of antibiotic-resistant bacteria in the Intensive Care Unit (ICU). More specifically, this project requires that a cluster-randomized trial (CRT) be designed and conducted to compare the effects of universal glove and gowning procedures as compared to the current standard of care in ICUs.

STUDY DESIGN: The study is a two arm, cluster-randomized trial. Randomization and analysis will be performed at the ICU level. A secondary statistical analysis will be performed at the patient level.

STUDY POPULATION: Adult patients in medical, surgical or combined medical/surgical ICUs.

SAMPLE SIZE: Based on the power calculations presented in Appendix I for each of the CRT aims, the study will use at least 18 ICU sites, half for the universal gown and glove intervention and half for CDC standards of care only. We will seek to maximize the number of ICUs involved to improve the scientific value of the study. The study is presently powered for a 1-year intervention study if 18 ICUs are included. After the 2 month pre-randomization period, we will use the actual number of sites enrolled and our baseline estimates to see if we can achieve the same degree of power for a study intervention of less than a year.

We have been able to recruit and retain 20 ICU sites. Upon completion of the pre-randomization period and based upon revised power calculations we will complete a 9-month intervention.

RANDOMIZATION: Randomization with pair matching based on the baseline data collection of outcomes will be used.

DATA ANALYSIS: Analyses of all aims will be performed according to the intention-to-treat (ITT) paradigm at the ICU level and will accommodate the matched-pairs design.

INTERVENTION:

Aim 1: Perform a CRT in which healthcare workers in the intervention ICUs will wear gloves and gowns for all patient contact while the control units perform regular standard and contact precautions per CDC guidelines in their respective ICUs.

Aim 1a: Measure the colonization acquisition rates of antibiotic-resistant pathogens in both intervention and non-intervention ICUs.

Aim 1b: Measure the HAI rates of catheter-associated bloodstream infection, catheter-associated urinary tract infection and ventilator-associated pneumonia in both intervention and non-intervention ICUs.

Aim 1c: Measure in-hospital 30-day mortality in both intervention and non-intervention ICUs.

Aim 1d: Measure hospital length of stay in both intervention and non-intervention ICUs.

Aim 1e: Measure the frequency of adverse events including frequency of healthcare worker visits and frequency of adverse events using an IHI adverse event tool.

Aim 1f: Statistically determine whether the intervention was effective in decreasing acquisition of antibiotic-resistant bacteria (primary outcome), reducing HAI rates (secondary outcome), decreasing in-hospital 30-day mortality (secondary outcome), decreasing length of stay (secondary outcome) and not increasing adverse events (secondary outcome).

HYPOTHESES:

Hypothesis 1a: Healthcare workers wearing gloves and gowns during all patient contact in the ICU setting will reduce antibiotic-resistant pathogen acquisition in at-risk patients.

Hypothesis 1b: Healthcare workers wearing gloves and gowns during all patient contact in the ICU setting will decrease HAI rates.

Hypothesis 1c: Healthcare workers wearing gloves and gowns during all patient contact in the ICU setting will decrease 30-day mortality.

Hypothesis 1d: Healthcare workers wearing gloves and gowns during all patient contact in the ICU setting will decrease hospital length of stay.

Hypothesis 1e: Healthcare workers wearing gloves and gowns during all patient contact in the ICU setting will not lead to an increase of adverse events.

CRITERIA FOR EVALUATION:

Primary Outcome:

The primary outcome of interest is the acquisition of an antibiotic-resistant pathogen, specifically Vancomycin-resistant Enterococcus (VRE) or Methicillin Resistant Staphylococcus Aureus(MRSA), as determined by peri-anal surveillance cultures for VRE and by nasal surveillance cultures for MRSA. The outcomes will be analyzed both individually and collectively (i.e., VRE, MRSA and VRE or MRSA).

Acquisition will be defined as:

1. A patient who has an initial ICU surveillance culture that is negative for an antibiotic-resistant pathogen and
2. Any subsequent surveillance culture within the same ICU admission that is positive for an antibiotic-resistant pathogen.

Secondary Outcomes:

The HAI rates to be measured will consist of catheter-associated bloodstream infection, catheter-associated urinary tract infection and ventilator-associated pneumonia rates. Hospital length of stay and 30-day mortality will also be measured as secondary outcomes. Adverse events are also a secondary outcome and will be measured using the frequency of healthcare worker visits and the frequency of adverse events as measured by an IHI tool.

ELIGIBILITY:
Inclusion Criteria:

ICUs to be included are: adult medical, surgical or combined medical surgical ICU as defined below:

* Medical ICU (MICU) > 80% of patients have a medical condition and have not undergone a surgical procedure during the current hospital stay
* Surgical ICU (SICU) > 80% of the patients have undergone a surgical procedure during the current hospital stay
* Combined Medical/Surgical ICU (MICU/SICU) - a roughly equivalent mixture of patients with medical conditions who have not undergone surgical procedures and patients who have undergone surgical procedures during the current hospital stay. Each group makes up > 20% and less than 80% of the total number of patients

  * Ability to collect the data required for analysis
  * Written approval of the study from the institution's IRB. The institution may opt to use the IRB approval provided by the centralized IRB at the University of Maryland, School of Medicine
  * Memorandum of Understanding signed by the ICU Medical Director, ICU Nurse Manager or Director and the Hospital Epidemiologist indicating a commitment to supporting enrollment of an ICU and completion the study
  * Ability to be matched with another ICU based on baseline acquisition of resistant bacteria on culture
  * Agreement to not perform active surveillance for MRSA or VRE that will be fed back to patients during the study period

Exclusion Criteria:

Pediatric ICUs and other non-medical or non-surgical ICUs will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients in medical, surgical or combined medical/surgical ICUs.
Sampling Method: Probability Sample
Enrollment: 19856 (Actual)
Dates: Start 2010-12; Primary Completion 2012-10-04 (Actual); Study Completion 2013-10-16 (Actual)

PRIMARY OUTCOMES:
Number of ICU Patients Who Acquire VRE or MRSA | 9 months
  The outcome of interest is the acquisition of VRE or MRSA as determined by peri-anal surveillance cultures for VRE and by nasal surveillance cultures for MRSA. The outcomes will be analyzed both individually and collectively.
  Acquisition will be defined as:
  1. A patient who has an initial ICU surveillance culture that is negative for an antibiotic-resistant pathogen.
  2. Subsequent discharge surveillance culture within the same ICU admission that is positive for an antibiotic-resistant pathogen.

SECONDARY OUTCOMES:
Number of ICU Patients Who Acquire CABSI | 9 months
  In all of the intensive-care units, catheter-associated bloodstream infection, catheter-associated urinary tract infection and ventilator-associated pneumonia rates will be measured in a standardized fashion at the cluster or group level. Data is collected on an individual patient basis in a de-identified fashion and will be reported to investigators at the cluster level
Number of ICU Patients Who Acquire CAUTI | 9 months
  In all of the intensive-care units, catheter-associated urinary tract infection rates will be measured in a standardized fashion at the cluster or group level. Data is collected on an individual patient basis in a de-identified fashion and will be reported to investigators at the cluster level
Number of ICU Patients Who Acquire VAP | 9 months
  In all of the intensive-care units, ventilator-associated pneumonia rates will be measured in a standardized fashion at the cluster or group level. Data is collected on an individual patient basis in a de-identified fashion and will be reported to investigators at the cluster level
Changes from Baseline in 30-day Mortality Rate | 9 months
  Thirty-day mortality will be a binary outcome of either the patient died at 30-days or was alive at 30-days after ICU admission date. This information will be recorded on an individual basis by the coordinator but will be reported on a group-level to the research center.
Changes from Baseline in ICU LOS | 9 months
  ICU length of stay will be a continuous variable. This information will be recorded on an individual basis by the coordinator but will be reported on a group-level to the research center.
Number of Adverse Events Occuring in the ICU | 9 months
  The study will look at a number of adverse events including 30-day mortality and the frequency of healthcare worker visits. Compliance with hand hygiene and the frequency of adverse events as measured by a modified Institute for Healthcare Improvement (IHI) trigger tool.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony D Harris, MD, MPH, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

REFERENCES:
- [Result] Harris AD, Pineles L, Belton B, Johnson JK, Shardell M, Loeb M, Newhouse R, Dembry L, Braun B, Perencevich EN, Hall KK, Morgan DJ; Benefits of Universal Glove and Gown (BUGG) Investigators; Shahryar SK, Price CS, Gadbaw JJ, Drees M, Kett DH, Munoz-Price LS, Jacob JT, Herwaldt LA, Sulis CA, Yokoe DS, Maragakis L, Lissauer ME, Zervos MJ, Warren DK, Carver RL, Anderson DJ, Calfee DP, Bowling JE, Safdar N. Universal glove and gown use and acquisition of antibiotic-resistant bacteria in the ICU: a randomized trial. JAMA. 2013 Oct 16;310(15):1571-80. doi: 10.1001/jama.2013.277815. PMID 24097234
- [Derived] Morgan DJ, Dubberke ER, Hink T, Paszkiewicz G, Burnham CD, Pineles L, Magder L, Johnson JK, Leekha S, Harris AD. The Impact of Universal Glove and Gown Use on Clostridioides Difficile Acquisition: A Cluster-Randomized Trial. Clin Infect Dis. 2023 Feb 8;76(3):e1202-e1207. doi: 10.1093/cid/ciac519. PMID 35776131
- [Derived] Harris AD, Morgan DJ, Pineles L, Magder L, O'Hara LM, Johnson JK. Acquisition of Antibiotic-Resistant Gram-negative Bacteria in the Benefits of Universal Glove and Gown (BUGG) Cluster Randomized Trial. Clin Infect Dis. 2021 Feb 1;72(3):431-437. doi: 10.1093/cid/ciaa071. PMID 31970393